CLINICAL TRIAL: NCT06452121
Title: Triglyceride-glucose Index as a Marker to Predict Severity of Coronary Artery Disease
Brief Title: TyG Index as a Marker to Predict Severity of Coronary Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Mohamed Mohsen Abdelaziz, Assistant Lecturer, Assiut University
Other Study IDs: TyG index and CAD
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
Keywords: triglyceride-glucose index
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients: to know severity of coronary artery disease using Triglyceride glucose (TyG) index in diabetic patients comparing it with non diabetic
  Interventions: Other: triglyceride glucose index
- Non diabetic patients: to know severity of coronary artery disease using Triglyceride glucose (TyG) index in non diabetic patients
  Interventions: Other: triglyceride glucose index

INTERVENTIONS:
Other: triglyceride glucose index — The TyG index was calculated using the following equation: Ln [TG (mg/dL)×FPG (mg/dL) / 2].
  CAD was referred to as at least one major coronary artery with≥50% stenosis evaluated by CAG

SUMMARY:
Triglyceride glucose (TyG) index is a novel marker, which has been demonstrated to have a high sensitivity and specificity in identifying metabolic syndrome . Previous studies have shown that TyG index is associated with carotid atherosclerosis, coronary artery calcification and high risk of CVD.

This study aims to predict severity of CAD using TyG index and its correlation to coronary angiography findings.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is characterized by vulnerable atherosclerotic plaque, which causes coronary stenosis and myocardial ischemia. The blockage of the blood vessel caused by the detachment of the endovascular plate leads to an acute CAD attack. Without timely intervention, this can be life-threatening for the patient. Currently, coronary angiography (CAG) is the reference standard for diagnosing CAD with inconclusive evidence to confirm the morbid state. Although it assesses the severity of coronary vascular occlusion, this technique is invasive and carries inherent risks.

Hypertriglyceridemia (HTG) is a common dyslipidemia and the association of triglyceride (TG) with CVD risk remains controversial . However, judging from a credible body of evidence, we can conclude that HTG is an independent risk factor of developing glucose metabolism disorders. Plasma TG levels are strongly associated with raised glucose levels because of the interactions between fat, muscle and function of pancreatic β-cells .

Moreover, accumulation of TG in the liver may cause fatty liver disease, which can increase the risk of type 2 diabetes mellitus (T2DM) . Prospective studies have revealed that plasma TG is an independent risk factor for developing T2DM . Additionally, it has been demonstrated that lowering TG, such as fibrates do, can significantly attenuate the process of developing insulin resistance . Furthermore, it also has been reported that both fasting glucose and TG within the high normal range may predict CVD risk . Hence, evaluating the joint value of TG and fasting glucose in patients with stable coronary artery disease (CAD) may be clinically in need.

Triglyceride glucose (TyG) index is a novel marker, which has been demonstrated to have a high sensitivity and specificity in identifying metabolic syndrome . Previous studies have shown that TyG index is associated with carotid atherosclerosis, coronary artery calcification and high risk of CVD.

Several studies demonstrated that the TyG index has a positive relevance with type 2 diabetes, Insulin resistence ,subclinical myocardial injury,and acute coronary syndrome (ACS). A higher TyG index correlates with a greater incidence of major adverse cardiovascular events in patients with diabetes and ACS, indicating its potential as an independent predictor for cardiovascular disease prognosis.

A recent large-scale prospective study suggested that the TyG index is an independent predictor for the progression of coronary artery calcification, especially in individuals without heavy coronary artery calcification at baseline . Moreover, an increased TyG index has been shown to be independently associated with higher risks of atherosclerotic cardiovascular diseases, including myocardial infarction, and worse prognosis in patients with ACS, irrespective of diabetes mellitus .

This study aims to predict severity of CAD using TyG index and its correlation to coronary angiography findings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above 18 years old presenting with either with ACS undergoing coronary angiography or Ischemic heart disease patients undergoing elective coronary angiography.

Exclusion Criteria:

* Pregnant or lactating women
* Patients with previous intravenous thrombolysis,
* Long -term use of statins or other lipid-regulating drugs
* Myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients above 18 years old presenting with either with ACS undergoing coronary angiography or Ischemic heart disease patients undergoing elective coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Predict severity of coronary artery disease change in Triglyceride glucose (TyG) index | cases during 1 year of the study
  Predict severity of coronary artery disease using Triglyceride glucose (TyG) index and its correlation to coronary angiography findings

CONTACTS AND LOCATIONS:
Overall Officials: Fatma M Abdelaziz, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geng X, Zhang X, Li X, Zhong C, Hou M. Triglyceride-glucose Index as a Valuable Marker to Predict Severity of Coronary Artery Disease: A Retrospective Cohort Study. Clin Appl Thromb Hemost. 2024 Jan-Dec;30:10760296241234320. doi: 10.1177/10760296241234320. PMID 38444211
- [Background] Jin JL, Cao YX, Wu LG, You XD, Guo YL, Wu NQ, Zhu CG, Gao Y, Dong QT, Zhang HW, Sun D, Liu G, Dong Q, Li JJ. Triglyceride glucose index for predicting cardiovascular outcomes in patients with coronary artery disease. J Thorac Dis. 2018 Nov;10(11):6137-6146. doi: 10.21037/jtd.2018.10.79. PMID 30622785